CLINICAL TRIAL: NCT02525757
Title: DETERRED: PD-L1 blockadE To Evaluate the Safety of Lung CanceR Therapy Using Carboplatin, Paclitaxel, and Radiation CombinEd With MPDL3280A
Brief Title: MPDL3280A With Chemoradiation for Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0722; NCI-2015-01543 (Registry Identifier: NCI-CTRP-Clinical Trial Reporting Registry)
Record Dates: First submitted 2015-08-14; First posted 2015-08-17 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Lung Cancer; Non-Small Cell Lung Cancer
Keywords: Lung Cancer; Non-small cell lung cancer; NSCLC; Unresectable; MPDL3280A; Carboplatin; Paraplatin; Paclitaxel; Taxol; Radiation therapy; XRT
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Carboplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Chemotherapy + Radiation (Experimental): Participants receive standard chemotherapy and radiation for 6-7 weeks, followed by a 3-4 week rest period when they receive no chemotherapy or radiation.
  Consolidation Phase: After the rest period, participants receive MPDL3280A in addition to chemotherapy for 2 cycles.
  Maintenance Phase: After completing the consolidation period, participants continue to receive MPDL3280A alone for up to 1 year.
  Interventions: Drug: MPDL3280A; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiation Therapy
- Group 2: MPDL3280A + Chemotherapy + Radiation (Experimental): Participants receive MPDL3280A, standard chemotherapy, and radiation therapy for 6-7 weeks. This will be followed by a rest period of 3-4 weeks, during which time participant receives 1 dose of MPDL3280A but no chemotherapy or radiation.
  Consolidation Phase: After the rest period, participants receive MPDL3280A in addition to chemotherapy for 2 cycles.
  Maintenance Phase: After completing the consolidation period, participants continue to receive MPDL3280A alone for up to 1 year.
  Interventions: Drug: MPDL3280A; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: MPDL3280A — 1200 mg by vein every 3 weeks up to 1 year after completing consolidation chemotherapy.
  Group 1: MPDL3280A given after receiving standard chemotherapy and radiation for 6-7 weeks, followed by a 3-4 week rest period.
  Group 2: MPDL3280A given with standard chemotherapy, and radiation therapy for 6-7 weeks followed by a rest period of 3-4 weeks, during which time participants receive 1 dose of MPDL3280A but no chemotherapy or radiation.
Drug: Carboplatin — AUC 2 by vein once a week on Day 1 during radiation therapy. During consolidation chemotherapy, Carboplatin given at AUC 6 by vein on Days 1 and 22 for 2 cycles.
  Other Names: Paraplatin
Drug: Paclitaxel — 50 mg/m2 by vein once a week on Day 1 during radiation therapy. During consolidation chemotherapy, Paclitaxel given at 200 mg/m2 on Days 1 and 22 for 2 cycles.
  Other Names: Taxol
Radiation: Radiation Therapy — 60-66 Gy in 30-33 fractions administered once-daily on Day 1, 5 days a week, for 6 to 7 weeks.
  Other Names: XRT

SUMMARY:
The goal of this clinical research study is to learn about the safety of adding MDPL3280A to standard chemotherapy (a combination of carboplatin and paclitaxel) and radiation in patients with lung cancer.

You are being asked to take part in this study because you have non-small cell lung cancer (NSCLC) that is unresectable (cannot be removed by surgery) and has not spread.

This is an investigational study. MPDL3280A is not FDA approved or commercially available. It is currently being used for research purposes only. Paclitaxel, carboplatin, and the radiation therapy are all FDA approved for the treatment of lung cancer. The use of these drugs in combination is considered investigational.

Up to 40 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Groups and Study Drug Administration:

Each study cycle is 21 days.

If you are found to be eligible to take part in this study, depending on when you join the study, you will be assigned to 1 of 2 study groups. Up to 10 participants will be assigned to Group 1 and up to 30 will be assigned to Group 2.

Participants in Groups 1 and 2 will receive standard chemotherapy 1 time each week and radiation therapy 5 days per week as described below Every cycle you will also receive MPDL3280A by vein over about 1 hour.

If you are in Group 1, you will receive standard chemotherapy and radiation for 6-7 weeks, followed by around a 3-8 week "rest period" when you will receive no chemotherapy or radiation.

If you are in Group 2, you will receive MPDL3280A, standard chemotherapy, and radiation therapy for 6-7 weeks. This will be followed by a rest period of 3-4 weeks, during which time you will receive 1 dose of MPDL3280A but no chemotherapy or radiation.

After the rest period, Groups 1 and 2 will both receive MPDL3280A in addition to chemotherapy for 2 cycles (called the consolidation period). After completing the consolidation period, you will continue to receive MPDL3280A alone for up to 1 year (called the maintenance period).

During your first dose of MPDL3280A, your vital signs (blood pressure, pulse, temperature, and breathing rate) will be measured 60 minutes before the dose, every 15 minutes during the dose, and 30 minutes after the dose to check for any bad reaction to the study drug. You may be given standard drugs to help with side effects.

If you need to stop receiving chemotherapy due to side effects, you will also stop receiving MPDL3280A. If you stop receiving chemotherapy for any other reason, you may continue receiving MPDL3280A.

Study Visits:

Once a week during Weeks 1-7:

* You will have a physical exam.
* Blood (up to 2 teaspoons) will be drawn for routine tests and to check your liver and kidney function.

Between Weeks 8-16 you will have a rest period. The rest period could range from 3-8 weeks, after which time you will return for the consolidation period.

One (1) time during consolidation period, which starts after the rest period, during Weeks 1-3 and Weeks 4-6 of the consolidation period:

* You will have a physical exam.
* Blood (up to 2 teaspoons) will be drawn for routine tests and to check your liver and kidney function.
* You will have either a CT scan or an FDG-PET/CT scan to check the status of the disease.

After you complete the consolidation period, you will enter the maintenance period. During every cycle of the maintenance period, blood (about 2 teaspoons) will be drawn for routine tests.

Every 2 cycles during the maintenance period, for up to 1 year:

* You will have a physical exam.
* You will have either a CT scan or an FDG-PET/CT scan to check the status of the disease.

If the disease appears to come back at any time during the study:

* You will have a physical exam.
* You will have a CT scan or MRI of the brain to check the status of the disease.
* You will have either a CT scan or an FDG-PET/CT of your chest and abdomen to check the status of the disease.
* You will have a biopsy of any suspicious areas found on the scans to check the status of the disease.
* Your doctor may choose to continue the study drug and repeat the scans in 6-8 weeks to check the status of the disease.
* If your doctor feels that the study drug is no longer effective from the information obtained from the repeat scans, you will be taken off the study drug. You will continue to be followed up by a schedule determined by your doctor.
* Your doctor may offer alternative treatments if your doctor feels it is in your best interest.

Length of Treatment:

You may receive the study drug for up to 1 year after starting the consolidation period, as long as the doctor thinks it is in your best interest. You will no longer be able to receive study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

If you are taken off study during the consolidation or maintenance period due to intolerable side effects, you will be followed by the study staff as often the doctor thinks is needed until the side effects get better.

Your active participation on the study will be over after the follow-up visits.

Follow-up Visits:

You will have follow-up visits every 2-4 months for up to 2 years after your last dose of study drug, unless you leave the study due to side effects or the disease having appeared to come back. After 2 years, you will have follow-up visits about every 4-6 months based on what your doctor thinks is best.

At each follow-up visit, the following tests will be performed:

* You will have a physical exam.
* You will have either a CT scan or an FDG-PET/CT scan of your chest and abdomen to check the status of the disease.
* If your doctor thinks it is needed, blood (up to 2 teaspoons) will be drawn for routine tests and to check your liver and kidney function.

If you cannot return to MD Anderson for these visits, you may be called by a member of the study staff every 3-6 months for 4 years after the last dose of study drug. Each call should last about 10 minutes. The study staff may ask that any tests or scans done by your home doctor be sent to MD Anderson to check the status of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to provide informed consent
2. Ability and willingness to comply with the requirements of the study protocol
3. Age >/= 18 years.
4. Representative tumor specimens in paraffin blocks (preferred) or at least 10 unstained slides, with an associated pathology report, requested at any time prior to study entry. Only tissue from core needle, punch, or excisional biopsy sample collection will be accepted. Fine-needle aspiration, brushing, and lavage samples are not acceptable. For all biopsy types, submitted blocks should have sufficient tissue to generate at least 10 sections, and tissue for which the pathology report specifies that the overall tumor content is low (e.g., "sparse" or "scant") is not acceptable.
5. Cont'd from #4: If archival tissue is either insufficient or unavailable, the patient will need to consent to and undergo a pre treatment core or excisional biopsy sample collection of the tumor. Fine needle aspiration, brushing, and lavage samples are not acceptable. The immediate unavailability of tissue blocks or unstained slides aside from the slides needed for diagnostic confirmation of lung cancer does not exclude patients from this trial. If the patient chooses to not undergo a repeat biopsy aside from biopsy for diagnostic purposes, the patient will still be eligible to enroll on 2014-0722. However, availability of core or excisional biopsy samples must be ascertained prior to enrollment.
6. Patients must have histologically confirmed, untreated non-small cell lung cancer that are considered non-metastatic, unresectable for which chemoradiation is the definitive therapy.
7. Patients will have the option to enroll on blood collection protocol, LAB09-0983, for serial collections of blood before, during intervals of treatment, and at follow up visits. Enrolling on the LAB09-0983 protocol is not required to enroll on the 2014-0722 study.
8. Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to the first study treatment (Cycle 1, Day 1): Absolute neutrophil count (ANC) >/= 1500 cells/uL *White Blood Cells (WBC) counts > 2500/uL *Lymphocyte count >/= 500/uL *Platelet count >/= 100,000/uL; for patients with hematologic malignancies, platelet count >/= 75,000/uL *Hemoglobin >/= 9.0 g/dL *Total bilirubin </= 1.5 x Upper Limit of Normal (ULN) with the following exception: Patients with known Gilbert disease who have serum bilirubin level </= 3 x ULN may be enrolled. *Aspartate Aminotransferase (AST) and Alanine transaminase (ALT) </= 3.0 x ULN
9. Cont'd from #8: Serum creatinine </= 1.5 x ULN or creatinine clearance >/= 50 mL/min on the basis of the Cockcroft-Gault glomerular filtration rate estimation: (140 - age) x (weight in kg) x (0.85 if female) / 72 x (serum creatinine in mg/dL)
10. Measurable disease per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1
11. For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use highly effective form(s) of contraception (i.e., one that results in a low failure rate [< 1% per year] when used consistently and correctly) and to continue its use for 12 months after the last dose of MPDL3280A, and for male patients continued use of contraception must be for a minimum of 3 months post-treatment.
12. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 as long as patients are eligible to receive chemotherapy along with concurrent radiotherapy
13. International Normalized (INR) and aPTT </= 1.5 x ULN * This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation (such as low-molecular weight heparin or warfarin) should be on a stable dose.

Exclusion Criteria:

1. Patients with any distant metastasis (liver, lung, bone, brain).
2. Any approved anticancer therapy, including chemotherapy, hormonal therapy, or radiotherapy, within 3 weeks prior to initiation of study treatment; however, the following are allowed: *Hormone-replacement therapy or oral contraceptives *Herbal therapy > 1 week prior to Cycle 1, Day 1 (herbal therapy intended as anticancer therapy must be discontinued at least 1 week prior to Cycle 1, Day 1)
3. Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, cirrhosis, fatty liver, and inherited liver disease
4. Patients with acute leukemias, accelerated/blast phase chronic myelogenous leukemia, chronic lymphocytic leukemia, Burkitt lymphoma, plasma cell leukemia, or non-secretory myeloma
5. Pregnancy, lactation, or breastfeeding
6. Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
7. Inability to comply with study and follow-up procedures
8. History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis *Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible. *Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible. *Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions: *Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations *Rash must cover less than 10% of body surface area (BSA)
9. Cont'd from #9: *Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%) *No acute exacerbations of underlying condition within the last 12 months (not requiring PUVA [psoralen plus ultraviolet A radiation], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high potency or oral steroids)
10. History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan
11. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
12. History of human immunodeficiency virus (HIV) infection or active hepatitis B (chronic or acute) or hepatitis C infection *Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible. *Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for hepatitis C virus ribonucleic acid (HCV RNA).
13. Active tuberculosis
14. Severe infections within 4 weeks prior to Cycle 1, Day 1 including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
15. Signs or symptoms of severe infection (sepsis) within 2 weeks prior to treatment start.
16. Major surgical procedure within 28 days prior to treatment start or anticipation of need for a major surgical procedure during the course of the study (EBUS and mediastinoscopy and VATS are not considered major surgical procedures).
17. Administration of a live, attenuated vaccine within 4 weeks before treatment start or anticipation that such a live attenuated vaccine will be required during the study *Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist) within 4 weeks prior to treatment start or at any time during the study.
18. Malignancies within 3 years prior to treatment start, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, or ductal carcinoma in situ treated surgically with curative intent) or undergoing active surveillance per standard-of-care management (e.g., CLL Rai Stage 0, prostate cancer with Gleason score </= 6, and PSA </= 10 mg/mL, etc.)
19. FOLLOWING ARE Medication-Related Exclusion Criteria: *Treatment with systemic immunostimulatory agents (including but not limited to IFN-a, IL-2) within 6 weeks or five half-lives of the drug (whichever is shorter) prior to the start of chemoradiation.Treatment with investigational agent within 4 weeks prior to Cycle 1, Day 1 (or within five half lives of the investigational product, whichever is longer)
20. Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents) within 2 weeks prior to Cycle 1, Day 1 *Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled. *The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
21. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
22. Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Time to Toxicity | 15 weeks
  Time to toxicity defined as any grade 3, 4 regimen-related non-hematologic toxicity, during the first 15 weeks of therapy. The method of Thall et al. used for safety monitoring.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 6 months and 1 year
  Six months and one year PFS is primary efficacy outcome measure. PFS defined as the freedom from any disease progression or death due to any cause. The 6 months benchmark is 75% and 1 year benchmark is 50% from the most recently completed trial RTOG 0617. PFS estimated by the inverse probability of treatment weighted (IPTW) Kaplan-Meier method [Robins et al., 2000; Cole et al., 2006].

CONTACTS AND LOCATIONS:
Overall Officials: Steven H. Lin, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Augustyn A, Adams DL, He J, Qiao Y, Verma V, Liao Z, Tang CM, Heymach JV, Tsao AS, Lin SH. Giant Circulating Cancer-Associated Macrophage-Like Cells Are Associated With Disease Recurrence and Survival in Non-Small-Cell Lung Cancer Treated With Chemoradiation and Atezolizumab. Clin Lung Cancer. 2021 May;22(3):e451-e465. doi: 10.1016/j.cllc.2020.06.016. Epub 2020 Jun 20. PMID 32798130
- See also: MD Anderson Cancer Center — http://www.mdanderson.org